CLINICAL TRIAL: NCT03055858
Title: AMPLATZER Duct Occluder II Additional Sizes Clinical Study
Brief Title: AMPLATZER Duct Occluder II Additional Sizes
Acronym: ADO II AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10171
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Patent Ductus Arteriosus
Keywords: PDA; SJM-CIP-10171; ADO II AS; IDE; CAP
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Intervention Model Description: ADO II AS device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- PDA closure (Experimental)
  Interventions: Device: ADO II AS (PDA closure)

INTERVENTIONS:
Device: ADO II AS (PDA closure) — Closure of PDA using Amplatzer Duct Occluder II Additional Sizes (ADO II AS).

SUMMARY:
The ADO II AS Study is a single arm, prospective, multicenter, nonrandomized clinical investigation to characterize the safety and effectiveness of the ADO II AS device in patients with a patent ductus arteriosus (PDA). Subjects will be implanted with the ADO II AS device using a transcatheter femoral vessel approach under fluoroscopic and echocardiographic guidance.

To account for subject dropout, up to 50 subjects will be enrolled in this clinical investigation. Up to an additional 150 subjects may be enrolled under continued access. The clinical investigation will be conducted at up to 10 centers in the United States.

Subjects participating in this clinical investigation will be followed for 3 years. The expected duration of enrollment is 18 months. The total duration of the clinical investigation is expected to be 4.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a PDA
* PDA ≤ 4mm in diameter
* PDA ≥ 3mm in length
* Subject (or legally authorized representative) is willing to comply with all pre-procedure, post-procedure, and follow-up testing requirements and provides consent to participate in the clinical study

NOTE: This study is enrolling children and all local laws and governing IRB requirements will be followed for obtaining informed consent

Exclusion Criteria:

* Weight < 700 grams at time of the procedure
* Age < 3 days at time of procedure
* Coarctation of the aorta
* Left pulmonary artery stenosis
* Cardiac output that is dependent on right to left shunt through the patent ductus arteriosus due to pulmonary hypertension
* Intracardiac thrombus
* Active infection requiring treatment at the time of implant
* Female subjects of child bearing potential are either pregnant or desire to become pregnant within six months post implant
* Other disease process likely to limit survival to less than six (6) months
* Participating in another study for an investigational drug and/or device that may clinically interfere with this study's endpoints

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Zahn, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (9):
- United States (9):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Arnold Palmer Hospital, Orlando, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Methodist LeBonheur Healthcare, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morray BH, Sathanandam SK, Forbes T, Gillespie M, Berman D, Armstrong AK, Shahanavaz S, Jones T, Rockefeller T, Justino H, Nykanen D, Weiler C, Gutfinger D, Zahn EM. 3-year follow-up of a prospective, multicenter study of the Amplatzer Piccolo Occluder for transcatheter patent ductus arteriosus closure in children >/= 700 grams. J Perinatol. 2023 Oct;43(10):1238-1244. doi: 10.1038/s41372-023-01741-1. Epub 2023 Aug 16. PMID 37587183
- [Derived] Sathanandam SK, Gutfinger D, O'Brien L, Forbes TJ, Gillespie MJ, Berman DP, Armstrong AK, Shahanavaz S, Jones TK, Morray BH, Rockefeller TA, Justino H, Nykanen DG, Zahn EM. Amplatzer Piccolo Occluder clinical trial for percutaneous closure of the patent ductus arteriosus in patients >/=700 grams. Catheter Cardiovasc Interv. 2020 Nov;96(6):1266-1276. doi: 10.1002/ccd.28973. Epub 2020 May 20. PMID 32433821

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 50 subjects were enrolled in the ADO II AS IDE study at 8 centers in the United States between 5 June 2017 and 25 January 2018. Following completion of enrollment in the IDE cohort, an additional 150 subjects were enrolled in the continued access protocol (CAP) between 26 March 2018 and 1 February 2019.
Period: Overall Study
Arm/Group | PDA Closure
Started | 200
IDE | 136
CAP | 46
Completed | 156
Not Completed | 44
Not completed — Death | 9
Not completed — Withdrawal by Subject | 11
Not completed — Lost to Follow-up | 6
Not completed — Missed Follow-Up Visits | 18

BASELINE CHARACTERISTICS:
Arm/Group | PDA Closure
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: The ADO II AS IDE study composed of 2 cohorts including IDE (n=50) and CAP (n=150)
  months
    IDE Cohort: number analyzed (Participants) | 50
    IDE Cohort | 16.37 (32.45)
    CAP Cohort: number analyzed (Participants) | 150
    CAP Cohort | 13.10 (34.23)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ADO II AS IDE study composed of 2 cohorts including IDE (n=50) and CAP (n=150)
  Participants
    IDE Cohort: number analyzed (Participants) | 50
    IDE Cohort: Female | 29
    IDE Cohort: Male | 21
    CAP Cohort: number analyzed (Participants) | 150
    CAP Cohort: Female | 69
    CAP Cohort: Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    IDE Cohort: number analyzed (Participants) | 50
    IDE Cohort: Hispanic or Latino | 1
    IDE Cohort: Not Hispanic or Latino | 44
    IDE Cohort: Unknown or Not Reported | 5
    CAP Cohort: number analyzed (Participants) | 150
    CAP Cohort: Hispanic or Latino | 16
    CAP Cohort: Not Hispanic or Latino | 129
    CAP Cohort: Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ADO II AS IDE study composed of 2 cohorts including IDE (n=50) and CAP (n=150)
  Participants
    IDE Cohort: number analyzed (Participants) | 50
    IDE Cohort: American Indian or Alaska Native | 0
    IDE Cohort: Asian | 0
    IDE Cohort: Native Hawaiian or Other Pacific Islander | 0
    IDE Cohort: Black or African American | 21
    IDE Cohort: White | 21
    IDE Cohort: More than one race | 0
    IDE Cohort: Unknown or Not Reported | 8
    CAP Cohort: number analyzed (Participants) | 150
    CAP Cohort: American Indian or Alaska Native | 1
    CAP Cohort: Asian | 10
    CAP Cohort: Native Hawaiian or Other Pacific Islander | 1
    CAP Cohort: Black or African American | 55
    CAP Cohort: White | 57
    CAP Cohort: More than one race | 5
    CAP Cohort: Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 200
PDA Length [Mean (Standard Deviation); unit: mm] — Population: The ADO II AS IDE study composed of 2 cohorts including IDE (n=50) and CAP (n=150)
  mm
    IDE: number analyzed (Participants) | 50
    IDE | 8.28 (2.70)
    CAP: number analyzed (Participants) | 150
    CAP | 9.51 (2.98)

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: The Rate of Major Complications After an Attempted ADO II AS Device Implant
Description: Major complications are defined as device (ADO II AS) or procedure-related adverse events resulting in any of the following:
  * death,
  * life-threatening adverse event,
  * persistent or significant disability/incapacity, and/or
  * a major open surgical intervention which is performed by a surgeon under general anesthesia
Time Frame: Through 180 days
Population: The ADO II AS IDE study composed of 2 cohorts including IDE (n=50) and CAP (n=150). The analysis population included the subjects who were available at the time of evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PDA Closure
Number analyzed (Participants) | 194
percentage of participants
  IDE Cohort: number analyzed (Participants) | 50
  IDE Cohort | 0 [0.00 to 7.11]
  CAP Cohort: number analyzed (Participants) | 144
  CAP Cohort | 2.8 [0.76 to 6.96]

2. Primary Outcome: Effectiveness Endpoint: The Rate of Effective Closure of the Ductus Arteriosus Among Subjects With a Successful ADO II AS Implant
Description: The primary effectiveness endpoint is the rate of effective closure of the ductus arteriosus among subjects with a successful ADO II AS implant as assessed by the presence of either a Grade 0 (none) or Grade 1 (trivial) shunt at the 6-month follow-up by transthoracic echocardiography (TTE).
Time Frame: At the 6-month follow-up
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PDA Closure
Number analyzed (Participants) | 173
percentage of participants
  IDE Cohort: number analyzed (Participants) | 44
  IDE Cohort | 100 [91.96 to 100.00]
  CAP Cohort: number analyzed (Participants) | 129
  CAP Cohort | 99.2 [95.76 to 99.98]

3. Secondary Outcome: The Rate of Significant Obstruction of the Pulmonary Artery or Aorta
Description: The rate of significant obstruction of the pulmonary artery or aorta through the 6-month follow-up visit per the following definitions:
  1. Significant obstruction of the left pulmonary artery is defined as less than 30% flow to the left lung by lung perfusion scan or a peak instantaneous gradient in left pulmonary artery ≥35 mmHg by echocardiogram if lung perfusion scan is not available. OR
  2. Significant obstruction of the aorta is defined as a gradient of ≥20 mmHg in the aortic isthmus by invasive aortic catheterization or a mean gradient ≥20 mmHg in the aortic isthmus by echocardiogram if invasive aortic catheterization is not available.
Time Frame: Through 6 month follow-up visit
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PDA Closure
Number analyzed (Participants) | 171
percentage of participants
  IDE Cohort: number analyzed (Participants) | 41
  IDE Cohort | 2.4 [0.06 to 12.86]
  CAP Cohort: number analyzed (Participants) | 130
  CAP Cohort | 0 [0.00 to 2.80]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PDA Closure
All-Cause Mortality (participants affected / at risk) | 9/200
Serious Adverse Events (participants affected / at risk) | 13/200
Other Adverse Events (participants affected / at risk) | 26/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PDA Closure (N=200)
Anemia (Blood and lymphatic system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Procedural Blood Loss (Injury, poisoning and procedural complications) | 1
Coarctation of Aorta (Cardiac disorders) | 1
Obstruction of The Aorta (Cardiac disorders) | 1
Pulmonary Hypertension (Blood and lymphatic system disorders) | 1
Death (General disorders) | 2
Desaturation (General disorders) | 1
Device Migration (Injury, poisoning and procedural complications) | 1
Death Related to Liver Failure and Chronic Lung Disease (General disorders) | 1
Progressive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Compromise (Respiratory, thoracic and mediastinal disorders) | 1
Necrotizing Enterocolitis (Gastrointestinal disorders) | 1
Bleeding (Blood and lymphatic system disorders) | 1
Device Embolization (Injury, poisoning and procedural complications) | 1
Stroke (Nervous system disorders) | 1
Left Vocal Cord Paralysis (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PDA Closure (N=200)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Device Embolization (Injury, poisoning and procedural complications) | 5
Fever (General disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Compromise (Respiratory, thoracic and mediastinal disorders) | 1
Anemia Requiring Transfusion (Blood and lymphatic system disorders) | 1
Hoarse Cry (General disorders) | 1
Tissue from Left Side of Atrial Septum (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
Hypotension (Blood and lymphatic system disorders) | 1
Infection (Infections and infestations) | 1
Obstruction of The Pulmonary Artery (Respiratory, thoracic and mediastinal disorders) | 2
Thrombus (Blood and lymphatic system disorders) | 1
Valve Damage (Cardiac disorders) | 1
Valvular Regurgitation (Cardiac disorders) | 5
Vascular Occlusion (Vascular disorders) | 2
Vessel Damage (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Deterioration in Resp Status (Respiratory, thoracic and mediastinal disorders) | 1
Right bundle branch block (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT03055858/Prot_SAP_001.pdf